CLINICAL TRIAL: NCT06210555
Title: Multiparametric MRI in a Prospective Cohort of Living Kidney Donors, Recipients, and Healthy Controls: Correlations With Markers of Renal Function, Fibrosis and Ageing
Acronym: MpRenal
Status: Recruiting | Type: Observational
Sponsor: Patrick Schjelderup (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Patrick Schjelderup, Principal Investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: Protocol_v2
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplantation; Multiparametric Magnetic Resonance Imaging; Living Donors; Renal Fibrosis; Senescence
Keywords: MRI; Multiparametric; Renal transplantation; Fibrosis; Kidney donor
MeSH Terms: conditions — Fibrosis | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Renal biopsies Blood- and urine: markers of renal ageing and fibrosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Living kidney donors: Living kidney donors
  Interventions: Procedure: Living kidney donation
- Transplant recipients: Recipients of kidneys from living donors
  Interventions: Procedure: Renal transplantation
- Healthy controls: Age- and sex matched healthy controls (Living kidney donors)

INTERVENTIONS:
Procedure: Renal transplantation — Operative procedure - receipt of a kidney
  Groups: Transplant recipients
Procedure: Living kidney donation — Operative procedure - donation of a kidney
  Groups: Living kidney donors

SUMMARY:
Development of renal fibrosis is the irreversible culmination of various renal diseases and independently predicts adverse outcomes. Currently renal fibrosis can only be diagnosed by performing a renal biopsy. The procedure is invasive and is limited by sampling bias.

In recent years there has been a significant development in magnetic resonance imaging (MRI) based techniques. MRI can provide highly detailed anatomical images. Other MRI measures allow quantitative measurements of perfusion, oxygenation, tissue stiffness and diffusion of water molecules within tissue. The combination of several MRI techniques sensitive to different biophysical tissue properties in a single scan session is referred to as multiparametric MRI (mpMRI).

Emerging evidence suggests that mpMRI could represent a method for indirect characterization of renal microstructure and extent of fibrosis. So far, studies performed in living kidney donors and recipients have been mostly cross-sectional. For mpMRI to transition to the clinical setting there is a need for validation of MRI-based measures with currently used reference methods for quantifying renal function and fibrosis.

The aim of this longitudinal observational study in a cohort of living kidney donors, recipients and healthy controls is to investigate the utility of repeated mpMRI over a period of 2 years. MRI-based measures will be compared to current reference methods for quantifying renal function and fibrosis.

The investigators hypothesize that there will be significant correlations between MRI-based measures, renal function determined by precise measurement of glomerular filtration rate and extent of fibrosis determined by renal biopsy. MRI-based measures are expected to be predictive of renal function decline and development of renal fibrosis.

This study could provide valuable data that will be helpful in moving the field of renal mpMRI forward, with the goal of providing a novel and non-invasive method for the diagnosis of renal pathology.

DETAILED DESCRIPTION:
Development of renal fibrosis is a characteristic end point of various renal diseases and independently predicts adverse renal outcomes. The most common cause of kidney allograft failure after 1 year is chronic allograft nephropathy which is characterized by interstitial fibrosis and tubular atrophy. At present the only method for quantifying renal fibrosis is a renal biopsy. Although the risk of complications is relatively low, the procedure is invasive, limiting its use for repeated assessments in a clinical setting. Furthermore, as only the renal cortex is usually sampled and because of the miniscule amount of tissue obtained there are issues of sampling bias and information on total renal fibrosis is limited. Estimated glomerular filtration rate (eGFR) is widely used for monitoring renal function but is insensitive for detecting allograft fibrosis.

Epidemiological data suggests that living kidney donors (LKD) are at increased risk of end stage renal disease compared to matched non-donors. Lower predonation renal function and higher age accentuate the risk. In a recent prospective study, renal cortex volume predicted renal outcome after 1 year in LKD.

In recent years there has been a rapid development in renal magnetic resonance imaging (MRI) techniques, allowing assessment of total renal morphology, microstructure, hemodynamics, oxygenation, and diffusion of water. Multiparametric MRI (mpMRI) refers to the combination of several MRI-based measures sensitive to different biophysical tissue properties in a single scan session. The information obtained could possibly provide a means of characterizing several aspects of renal function and morphology.

The MRI based measures that show the greatest promise for clinical application are longitudinal relaxation time (T1), diffusion weighted imaging (DWI), blood oxygen-level dependent imaging (BOLD) and arterial spin labelling (ASL). In a cross-sectional study, patients with chronic kidney disease (n=22) and healthy volunteers (n=22) were assessed with MRI-based measures and renal biopsy. MRI based measures were reproducible and correlated with currently used methods for measuring renal function. Significant differences were found in T1-mapping, apparent diffusion coefficient (ADC) and ASL in persons with low and high degrees of renal fibrosis. In another cross-sectional study (n = 164) the corticomedullary ADC difference was highly correlated to and independently associated with renal fibrosis in both native kidneys and allografts. In a more recent prospective study, the corticomedullary ADC difference was predictive of kidney function decline and dialysis initiation in transplant recipients and patients with CKD. Reduced oxygenation determined by low BOLD has been linked to the progression rate of chronic kidney disease. Interestingly, a study found that diffusion-based MRI measures detected an increase in allograft fibrosis before apparent changes in the estimated glomerular filtration rate.

Before mpMRI of the kidneys can be utilized in the clinical setting there is a need for development of a larger evidence base. To date clinical studies employing MRI-based measures have been mostly cross-sectional. So far, only few studies have been performed in living kidney donors (LKD) and renal transplant recipients. To the best of our knowledge, no studies have been performed with long term follow-up including repeated mpMRI, renal biopsies and accurate measurement of glomerular filtration rate with DTPA clearance. Repeated imaging is necessary to establish how MRI-based measures change over time in association with currently used reference methods for quantifying renal function and fibrosis.

Accelerated renal ageing trough p16INK4a pathway activation, leading to cellular senescence, is involved in the development of renal fibrosis. Senescent cells are characterized by irreversible growth arrest and express a pro-inflammatory and pro-fibrotic senescent associated secretory phenotype (SASP). This biochemical footprint can be detected by immunohistochemistry and may be predictive of renal fibrosis in chronic kidney disease and renal transplantation.

Serum uromodulin (sUmod) and urinary epidermal growth factor (uEGF) originate from kidney tubules and may reflect functional nephron mass and are associated with renal function decline and fibrosis.

Klotho, which was initially known as an anti-ageing gene is expressed on the cell surface membranes of proximal and distal tubules. Decreasing levels of soluble klotho accompany chronic kidney disease and have been linked to the development of renal fibrosis.

The overall aim of this prospective follow-up study is to investigate the utility of repeated mpMRI and biomarkers in monitoring renal function and for detecting the development of fibrosis in renal allografts. MRI-based measures and biomarkers of renal ageing and fibrosis will be compared to current gold standard methods for characterizing and quantifying renal function and fibrosis in a cohort of LKD, recipients and healthy controls.

This is an exploratory study. A novel and unstandardized MRI patch consisting of multiple MRI-based measures performed in a single scan will be utilized. Specific data to inform estimates of accuracy and variance for this method is not available. Calculations of power and sample size are thus challenging to perform. Furthermore, published data on the relationships between MRI-based measures and fibrosis are heterogenous regarding the methods used for quantifying fibrosis histologically and thresholds for fibrosis.

The prevalence of fibrosis in renal allografts, which is of primary interest is expected to increase from baseline to the final visit. Based on previous work it is expected that 40-50 % of renal allografts will have significant levels of fibrosis after 2 years. It is however possible, that present levels of fibrosis in allografts are lower than previous due to optimized immunosuppressive regimens.

Several power calculations have been performed. Effect sizes have been based on prior published data on the difference and variance of ASL and ADC values in patients with different levels of fibrosis. With a power of 0.8 and an alpha of 0.05 it is estimated that a sample size n = 32 will be adequate to detect fibrosis at a threshold of 40%.

During the inclusion period LKD and recipients from Aalborg- and Aarhus University Hospital will be offered to participate in the study. Currently approximately 30-35 living donor pairs are transplanted annually. During the inclusion period of 2 years, the investigators aim to include 40 living donors and recipients. With an expected drop-out of 20% 32 living donors and recipients are expected to complete the study.

Multiparametric MRI mpMRI will be performed according to standard operating procedure in the Department of Diagnostic imaging at the participating hospitals.

The mpMRI scan protocol will be performed on a 3 Tesla MRI scanner (General Electrics (GE) Healthcare) and includes the following MRI measures:

* Structural T2 and/or T1 weighted renal MRI (for volumetric measurement)
* Diffusion weighted imaging (DWI) with b-values 0, 10, 20, 30, 40, 50, 70, 100, 200, 300, 400, 500, 800 s/mm2
* T1- and T2-mapping
* BOLD MRI with T2*
* ASL perfusion
* Non-contrast Magnetic Resonance Angiography
* Quantitative flow measurements in the renal arteries

Scan time is approximately 60 minutes. During this time participants will be required to lie still in the supine position. Participants will be required to fast for 3 hours prior to the scan.

Postprocessing of MRI data will be done with the aid of commercially available software and analysis software developed in-house in collaboration with Aalborg- and Aarhus University Hospital and Aarhus university.

99mTc-DTPA clearance is a method for accurately measuring GFR. The DTPA clearance will be performed according to standard operating procedure at the Departments of Diagnostic Imaging at the participating hospitals.

Allograft biopsy Biopsies will be obtained using 18G needle and fixed in phosphate-buffered 4% formaldehyde and embedded in paraffin and stained with hematoxylin and eosin, periodic acid-Schiff, and Masson trichrome.

Quantitative histological evaluation will be used to evaluate biopsies using and Olympus BX50 light microscope (Olympus Denmark, Ballerup, Denmark) equipped with a prior motorized stage, and Olympus DP70 digital camera interfaced to a PC with commercially available newCAST software (Visiopharm, Hørsholm, Denmark).

Extent of fibrosis will be quantified by systematic evaluation of scattered test points (≈100) across the Masson trichrome-stained sections using a x4 lens (NA 0.13) (29).

Additionally, biopsies will be evaluated for markers of renal ageing and fibrosis:

* p16INK4a pathway activation
* klotho
* additional markers of renal ageing and fibrosis

Blood- and urine samples Hemoglobin, hematocrit, leukocytes, platelets, CRP, creatinine, eGFR, urea, sodium, potassium, total phosphate, bicarbonate, ionized calcium, total magnesium, intact PTH, alkaline phosphatase, glucose, soluble klotho and sUmod.

A spot urine sample will be used for the determination of u-albumin/creatinine ratio, glucose, leucocytes, nitrite, blood and uEGF.

ELIGIBILITY:
Living kidney donors and transplant recipients:

Inclusion Criteria:

* Approved as a living kidney donor or recipient of a kidney from a living donor.
* Able to cooperate to an MRI examination

Exclusion Criteria:

* Contraindications to MRI due to incompatible foreign objects.
* Severe claustrophobia

Healthy controls:

Inclusion Criteria:

* Office BP < 140/90 mmHg. (use of 1 antihypertensive drug allowed)
* Normal eGFR. (CKD-EPI)
* Urine albumin-to-creatinine ratio < 30 mg/g.
* Dipstick negative for hematuria and proteinuria.
* Able to cooperate to an MRI examination.

Exclusion Criteria:

* Contraindications to MRI due to incompatible foreign objects.
* Severe claustrophobia.
* Pregnancy.
* Condition(s) that would exclude living kidney donation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective cohort of living kidney donors, recipients and healthy controls. Donors and recipients will be recruited from the Departments of Renal Medicine at Aalborg- and Aarhus University Hospital. Healthy controls will be matched by age and sex to living kidney donors.
  Based on power calculations we aim to include 32 participants in each cohort. Inclusion period of 2 years is expected and 2 years of follow-up planned.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between MRI-based measures (T1/T2-mapping, ADC, ASL) and fibrosis quantified by morphometric evaluation renal biopsy. | Multiparametric MRI and allograft biopsy at baseline, 3 months, 12 months and 24 months.
  Changes in MRI-based measures will be correlated to changes in allograft fibrosis quantified by morphometric evaluation of renal biopsy.

SECONDARY OUTCOMES:
Correlation between MRI-based measures (T1/T2-mapping, ADC, ASL) and measured GFR. | Multiparametric MRI and DTPA clearance baseline, 3 months, 12 months and 24 months.
  Changes in MRI-based measures will be correlated to changes in measured GFR. (DTPA clearance)
Diagnostic performance of MRI-based measures and biomarkers as regards to allograft fibrosis. | Multiparametric MRI and biomarkers at baseline, 3 months, 12 months and 24 months.
  Receiver operating characteristic curves, sensitivity, specificity, positive- and negative predicitive values will be specified.
Predictive value of MRI-based measures and biomarkers of renal ageing and fibrosis as regards to development of allograft fibrosis and renal function decline. | Multiparametric MRI and biomarkers at baseline, 3 months, 12 months and 24 months.
  Multiple regression modelling with MRI-based measures and biomarkers as independent variables and measured GFR and allograft fibrosis as dependent variables.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schjelderup, MD, Principal Investigator — Aalborg University Hospital
Locations (2):
- Denmark (2):
  - Department of Renal Medicine, Aarhus University Hospital, Aarhus, Central Jutland
  - Department of Nephrology, Aalborg University Hospital, Aalborg, North Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nath KA. Tubulointerstitial changes as a major determinant in the progression of renal damage. Am J Kidney Dis. 1992 Jul;20(1):1-17. doi: 10.1016/s0272-6386(12)80312-x. PMID 1621674
- [Background] Eknoyan G, McDonald MA, Appel D, Truong LD. Chronic tubulo-interstitial nephritis: correlation between structural and functional findings. Kidney Int. 1990 Oct;38(4):736-43. doi: 10.1038/ki.1990.266. No abstract available. PMID 2232511
- [Background] Park WD, Griffin MD, Cornell LD, Cosio FG, Stegall MD. Fibrosis with inflammation at one year predicts transplant functional decline. J Am Soc Nephrol. 2010 Nov;21(11):1987-97. doi: 10.1681/ASN.2010010049. Epub 2010 Sep 2. PMID 20813870
- [Background] Vadivel N, Tullius SG, Chandraker A. Chronic allograft nephropathy. Semin Nephrol. 2007 Jul;27(4):414-29. doi: 10.1016/j.semnephrol.2007.03.004. PMID 17616274
- [Background] Uslu A, Hur E, Sen C, Sen S, Akgun A, Tasli FA, Nart A, Yilmaz M, Toz H. To what extent estimated or measured GFR could predict subclinical graft fibrosis: a comparative prospective study with protocol biopsies. Transpl Int. 2015 May;28(5):575-81. doi: 10.1111/tri.12534. Epub 2015 Feb 27. PMID 25639483
- [Background] Mjoen G, Hallan S, Hartmann A, Foss A, Midtvedt K, Oyen O, Reisaeter A, Pfeffer P, Jenssen T, Leivestad T, Line PD, Ovrehus M, Dale DO, Pihlstrom H, Holme I, Dekker FW, Holdaas H. Long-term risks for kidney donors. Kidney Int. 2014 Jul;86(1):162-7. doi: 10.1038/ki.2013.460. Epub 2013 Nov 27. PMID 24284516
- [Background] O'Keeffe LM, Ramond A, Oliver-Williams C, Willeit P, Paige E, Trotter P, Evans J, Wadstrom J, Nicholson M, Collett D, Di Angelantonio E. Mid- and Long-Term Health Risks in Living Kidney Donors: A Systematic Review and Meta-analysis. Ann Intern Med. 2018 Feb 20;168(4):276-284. doi: 10.7326/M17-1235. Epub 2018 Jan 30. PMID 29379948
- [Background] Buus NH, Nielsen CM, Skov K, Ibsen L, Krag S, Nyengaard JR. Prediction of Renal Function in Living Kidney Donors and Recipients of Living Donor Kidneys Using Quantitative Histology. Transplantation. 2023 Jan 1;107(1):264-273. doi: 10.1097/TP.0000000000004266. Epub 2022 Jul 27. PMID 35883240
- [Background] Cox EF, Buchanan CE, Bradley CR, Prestwich B, Mahmoud H, Taal M, Selby NM, Francis ST. Multiparametric Renal Magnetic Resonance Imaging: Validation, Interventions, and Alterations in Chronic Kidney Disease. Front Physiol. 2017 Sep 14;8:696. doi: 10.3389/fphys.2017.00696. eCollection 2017. PMID 28959212
- [Background] Caroli A, Pruijm M, Burnier M, Selby NM. Functional magnetic resonance imaging of the kidneys: where do we stand? The perspective of the European COST Action PARENCHIMA. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii1-ii3. doi: 10.1093/ndt/gfy181. No abstract available. PMID 30137582
- [Background] Simms R, Sourbron S. Recent findings on the clinical utility of renal magnetic resonance imaging biomarkers. Nephrol Dial Transplant. 2020 Jun 1;35(6):915-919. doi: 10.1093/ndt/gfaa125. No abstract available. PMID 32516808
- [Background] Francis ST, Selby NM, Taal MW. Magnetic Resonance Imaging to Evaluate Kidney Structure, Function, and Pathology: Moving Toward Clinical Application. Am J Kidney Dis. 2023 Oct;82(4):491-504. doi: 10.1053/j.ajkd.2023.02.007. Epub 2023 May 13. PMID 37187282
- [Background] Buchanan CE, Mahmoud H, Cox EF, McCulloch T, Prestwich BL, Taal MW, Selby NM, Francis ST. Quantitative assessment of renal structural and functional changes in chronic kidney disease using multi-parametric magnetic resonance imaging. Nephrol Dial Transplant. 2020 Jun 1;35(6):955-964. doi: 10.1093/ndt/gfz129. PMID 31257440
- [Background] Berchtold L, Friedli I, Crowe LA, Martinez C, Moll S, Hadaya K, de Perrot T, Combescure C, Martin PY, Vallee JP, de Seigneux S. Validation of the corticomedullary difference in magnetic resonance imaging-derived apparent diffusion coefficient for kidney fibrosis detection: a cross-sectional study. Nephrol Dial Transplant. 2020 Jun 1;35(6):937-945. doi: 10.1093/ndt/gfy389. PMID 30608554
- [Background] Sugiyama K, Inoue T, Kozawa E, Ishikawa M, Shimada A, Kobayashi N, Tanaka J, Okada H. Reduced oxygenation but not fibrosis defined by functional magnetic resonance imaging predicts the long-term progression of chronic kidney disease. Nephrol Dial Transplant. 2020 Jun 1;35(6):964-970. doi: 10.1093/ndt/gfy324. PMID 30418615
- [Background] Berchtold L, Crowe LA, Friedli I, Legouis D, Moll S, de Perrot T, Martin PY, Vallee JP, de Seigneux S. Diffusion magnetic resonance imaging detects an increase in interstitial fibrosis earlier than the decline of renal function. Nephrol Dial Transplant. 2020 Jul 1;35(7):1274-1276. doi: 10.1093/ndt/gfaa007. No abstract available. PMID 32160279
- [Background] Selby NM, Blankestijn PJ, Boor P, Combe C, Eckardt KU, Eikefjord E, Garcia-Fernandez N, Golay X, Gordon I, Grenier N, Hockings PD, Jensen JD, Joles JA, Kalra PA, Kramer BK, Mark PB, Mendichovszky IA, Nikolic O, Odudu A, Ong ACM, Ortiz A, Pruijm M, Remuzzi G, Rorvik J, de Seigneux S, Simms RJ, Slatinska J, Summers P, Taal MW, Thoeny HC, Vallee JP, Wolf M, Caroli A, Sourbron S. Magnetic resonance imaging biomarkers for chronic kidney disease: a position paper from the European Cooperation in Science and Technology Action PARENCHIMA. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii4-ii14. doi: 10.1093/ndt/gfy152. PMID 30137584
- [Background] Docherty MH, O'Sullivan ED, Bonventre JV, Ferenbach DA. Cellular Senescence in the Kidney. J Am Soc Nephrol. 2019 May;30(5):726-736. doi: 10.1681/ASN.2018121251. Epub 2019 Apr 18. PMID 31000567
- [Background] van Deursen JM. The role of senescent cells in ageing. Nature. 2014 May 22;509(7501):439-46. doi: 10.1038/nature13193. PMID 24848057
- [Background] Melk A, Schmidt BM, Vongwiwatana A, Rayner DC, Halloran PF. Increased expression of senescence-associated cell cycle inhibitor p16INK4a in deteriorating renal transplants and diseased native kidney. Am J Transplant. 2005 Jun;5(6):1375-82. doi: 10.1111/j.1600-6143.2005.00846.x. PMID 15888044
- [Background] Chan J, Svensson M, Tannaes TM, Waldum-Grevbo B, Jenssen T, Eide IA. Associations of Serum Uromodulin and Urinary Epidermal Growth Factor with Measured Glomerular Filtration Rate and Interstitial Fibrosis in Kidney Transplantation. Am J Nephrol. 2022;53(2-3):108-117. doi: 10.1159/000521757. Epub 2022 Feb 1. PMID 35104815
- [Background] Yepes-Calderon M, Sotomayor CG, Kretzler M, Gans ROB, Berger SP, Navis GJ, Ju W, Bakker SJL. Urinary Epidermal Growth Factor/Creatinine Ratio and Graft Failure in Renal Transplant Recipients: A Prospective Cohort Study. J Clin Med. 2019 Oct 13;8(10):1673. doi: 10.3390/jcm8101673. PMID 31614925
- [Background] Kottgen A, Hwang SJ, Larson MG, Van Eyk JE, Fu Q, Benjamin EJ, Dehghan A, Glazer NL, Kao WH, Harris TB, Gudnason V, Shlipak MG, Yang Q, Coresh J, Levy D, Fox CS. Uromodulin levels associate with a common UMOD variant and risk for incident CKD. J Am Soc Nephrol. 2010 Feb;21(2):337-44. doi: 10.1681/ASN.2009070725. Epub 2009 Dec 3. PMID 19959715
- [Background] Scherberich JE, Gruber R, Nockher WA, Christensen EI, Schmitt H, Herbst V, Block M, Kaden J, Schlumberger W. Serum uromodulin-a marker of kidney function and renal parenchymal integrity. Nephrol Dial Transplant. 2018 Feb 1;33(2):284-295. doi: 10.1093/ndt/gfw422. PMID 28206617
- [Background] Cho NJ, Han DJ, Lee JH, Jang SH, Kang JS, Gil HW, Park S, Lee EY. Soluble klotho as a marker of renal fibrosis and podocyte injuries in human kidneys. PLoS One. 2018 Mar 28;13(3):e0194617. doi: 10.1371/journal.pone.0194617. eCollection 2018. PMID 29590173
- [Background] Buchanan S, Combet E, Stenvinkel P, Shiels PG. Klotho, Aging, and the Failing Kidney. Front Endocrinol (Lausanne). 2020 Aug 27;11:560. doi: 10.3389/fendo.2020.00560. eCollection 2020. PMID 32982966
- [Background] Nankivell BJ, Borrows RJ, Fung CL, O'Connell PJ, Allen RD, Chapman JR. The natural history of chronic allograft nephropathy. N Engl J Med. 2003 Dec 11;349(24):2326-33. doi: 10.1056/NEJMoa020009. PMID 14668458
- [Background] Stegall MD, Park WD, Larson TS, Gloor JM, Cornell LD, Sethi S, Dean PG, Prieto M, Amer H, Textor S, Schwab T, Cosio FG. The histology of solitary renal allografts at 1 and 5 years after transplantation. Am J Transplant. 2011 Apr;11(4):698-707. doi: 10.1111/j.1600-6143.2010.03312.x. Epub 2010 Nov 9. PMID 21062418